CLINICAL TRIAL: NCT03710772
Title: A Phase II Study of Ibrutinib Plus Rituximab Followed by Venetoclax and Hyper-CVAD Consolidation in Newly Diagnosed Young Patients With Mantle Cell Lymphoma: Window II Protocol
Brief Title: Ibrutinib, Rituximab, Venetoclax, and Combination Chemotherapy in Treating Patients With Newly Diagnosed Mantle Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0447; NCI-2018-02137 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0447 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-10-15; First posted 2018-10-18 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Cyclophosphamide; Cytarabine; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Doxorubicin; ibrutinib; Methotrexate; merphos; Rituximab; CT-P10; venetoclax; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group I (ibrutinib, rituximab, venetoclax, chemotherapy) (Experimental): Patients receive ibrutinib, rituximab, and venetoclax as described in part I.
  COMBINATION CHEMOTHERAPY: Patients receive rituximab IV over 6 hours on day 1, dexamethasone PO or IV on days 1-4, cyclophosphamide IV over 3 hours BID on days 2-4, and doxorubicin hydrochloride IV over 24 hours and vincristine sulfate IV over 15-30 minutes on day 5 of odd-numbered cycles (1 and 3). Patients also receive rituximab IV over 6 hours on day 1, methotrexate IV over 24 hours on day 2, and cytarabine IV over 2 hours BID on days 3-4 of even-numbered cycles (2 and 4). Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive ibrutinib and venetoclax PO QD on days 1-28, and rituximab IV over 4-8 hours on day 1 of every other month. Cycles repeat every 28 days for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Ibrutinib; Drug: Methotrexate; Biological: Rituximab; Drug: Venetoclax; Drug: Vincristine Sulfate
- Group II (ibrutinib, rituximab, venetoclax, chemotherapy) (Experimental): Patients receive ibrutinib, rituximab, and venetoclax as in part I.
  Patients receive combination chemotherapy as in group I. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive maintenance therapy as in group I.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Ibrutinib; Drug: Methotrexate; Biological: Rituximab; Drug: Venetoclax; Drug: Vincristine Sulfate
- Group III (ibrutinib, rituximab, venetoclax) (Experimental): Patients receive ibrutinib, rituximab, venetoclax as in part I. Patients then receive maintenance therapy as in group I.
  Interventions: Drug: Ibrutinib; Biological: Rituximab; Drug: Venetoclax

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
  Arms: Group I (ibrutinib, rituximab, venetoclax, chemotherapy); Group II (ibrutinib, rituximab, venetoclax, chemotherapy)
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
  Arms: Group I (ibrutinib, rituximab, venetoclax, chemotherapy); Group II (ibrutinib, rituximab, venetoclax, chemotherapy)
Drug: Dexamethasone — Given PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
  Arms: Group I (ibrutinib, rituximab, venetoclax, chemotherapy); Group II (ibrutinib, rituximab, venetoclax, chemotherapy)
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
  Arms: Group I (ibrutinib, rituximab, venetoclax, chemotherapy); Group II (ibrutinib, rituximab, venetoclax, chemotherapy)
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
  Arms: Group I (ibrutinib, rituximab, venetoclax, chemotherapy); Group II (ibrutinib, rituximab, venetoclax, chemotherapy)
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate
  Arms: Group I (ibrutinib, rituximab, venetoclax, chemotherapy); Group II (ibrutinib, rituximab, venetoclax, chemotherapy)

SUMMARY:
This phase II trial studies how well ibrutinib and rituximab given together with venetoclax and combination chemotherapy work in treating patients with newly diagnosed mantle cell lymphoma. Ibrutinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Rituximab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Venetoclax may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Drugs used in chemotherapy such as, cyclophosphamide, vincristine, doxorubicin, and dexamethasone, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving ibrutinib, rituximab, and venetoclax together with combination chemotherapy may work better in treating patients with mantle cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the complete response rate of the ibrutinib plus rituximab combination followed by venetoclax in newly diagnosed young mantle cell lymphoma (MCL) patients.

SECONDARY OBJECTIVES:

I. To determine the safety profile of the ibrutinib plus rituximab combination followed by venetoclax in newly diagnosed young MCL patients.

II. To evaluate the progression-free survival and overall survival time of the ibrutinib plus rituximab combination followed by venetoclax and hyper-fractionated cyclophosphamide, vincristine sulfate, doxorubicin hydrochloride, and dexamethasone (hyper-CVAD) in newly diagnosed young MCL patients.

EXPLORATORY OBJECTIVE:

I. Developing a novel biomarker for minimal residual disease (MRD) assay using the circulating tumor deoxyribonucleic acid (DNA) (ctDNA) assay on a customized capture sequencing gene panel for MCL using serial plasma samples collected in this trial.

OUTLINE:

PART I: Patients receive ibrutinib orally (PO) once daily (QD) on days 1-28 and receive rituximab intravenously (IV) over 4-8 hours on days 1, 8, 15, and 22 of cycle 1 and on day 1 of cycles 3-12. Patients also receive venetoclax PO QD on days 1-28 of cycles 5-12. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

PART II: Patients are assigned to 1 of 3 groups depending on risk status.

GROUP I:

COMBINATION CHEMOTHERAPY: Patients receive rituximab IV over 6 hours on day 1, dexamethasone PO or IV on days 1-4, cyclophosphamide IV over 3 hours twice daily (BID) on days 2-4, and doxorubicin hydrochloride IV over 24 hours and vincristine sulfate IV over 15-30 minutes on day 5 of odd-numbered cycles (1 and 3). Patients also receive rituximab IV over 6 hours on day 1, methotrexate IV over 24 hours on day 2, and cytarabine IV over 2 hours BID on days 3-4 of even-numbered cycles (2 and 4). Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Patients receive ibrutinib and venetoclax PO QD on days 1-28, and rituximab IV over 4-8 hours on day 1 of every other month. Cycles repeat every 28 days for up to 24 months in the absence of disease progression or unacceptable toxicity.

GROUP II: Patients receive combination chemotherapy as in group I. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive maintenance therapy as in group I.

GROUP III: Patients receive maintenance therapy as in group I.

After completion of study treatment, patients are followed up at 30 days, every 4 months for 2 years, every 6 months for 2 years, and then annually for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of mantle cell lymphoma with CD20 positivity in tissue biopsy
* MCL patients must have a clinical indication to start systemic therapy. Symptoms and features of MCL include any of the following: a) B-symptoms, b) Mantle Cell Lymphoma International Prognostic Index (MIPI) > 3, c) Ki 67 >= 30%, d) bulky tumors > 10 cm or in case of >= 2 tumors, each >= 5 cm in diameter, e) disease threatening organ function, f) elevated lactate dehydrogenase (LDH), g) peripheral blood (PB) white blood cell (WBC) > 50,000, h) pancytopenia due to bone marrow MCL, i) patient's choice due to anxiety; j) pain due to lymphoma; k) somatic mutations in the TP53, NSD2 or NOTCH genes; l) size of spleen >= 20 cm
* Newly diagnosed MCL with no prior therapy
* Sign (or their legally-acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study
* Bi-dimensional measurable disease using both computed tomography (CT) scan and/or positron emission tomography (PET)-CT or gastrointestinal biopsies, CT gastrointestinal, bone marrow or spleen only patients are allowable
* Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less
* Absolute neutrophil count (ANC) >= 1000/mm^3 independent of growth factor support
* Platelets >= 100,000/mm^3 or >= 50,000/mm^3 if bone marrow involvement without necessitating transfusion
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x upper limit of normal (ULN)
* Total bilirubin =< 1.5 x ULN unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin
* Creatinine clearance (CLcr) > 50 mL/min
* Cardiac ejection fraction >= 50% by echocardiogram (ECHO) or multigated acquisition (MUGA)
* Disease free of prior malignancies with exception of currently treated basal cell, squamous cell carcinoma of the skin, carcinoma "in situ" of the cervix or breast, or other malignancies in remission (including prostate cancer patients in remission from radiation therapy, surgery or brachytherapy), not actively being treated with life expectancy of greater than 3 years. Principal investigator (PI) can use clinical judgement in the best interest of patients
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test (within 28 days of initiation of protocol therapy) and must be willing to use acceptable methods of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials. Men must agree to use a latex condom during sexual contact with a female of childbearing potential even if they have had a successful vasectomy. Men must agree to not donate sperm during and after the study. For females, these restrictions apply for 1 month after the last dose of study drug. For males, these restrictions apply for 3 months after the last dose of study drug

  * A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

Exclusion Criteria:

* Any serious medical condition including but not limited to, uncontrolled hypertension, uncontrolled diabetes mellitus, active/symptomatic coronary artery disease, chronic obstructive pulmonary disease (COPD), renal failure, active hemorrhage, laboratory abnormality, or psychiatric illness that, in the investigators opinion, places the patient at unacceptable risk or would prevent the subject from signing the informed consent form
* Pregnant or breast-feeding females
* Known human immunodeficiency virus (HIV) infection (HIV testing is not required)
* Evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

  * Uncontrolled and/or active systemic infection (viral, bacterial or fungal)
  * Chronic hepatitis B virus (HBV) or hepatitis C (HCV) requiring treatment. Note: subjects with serologic evidence of prior vaccination to HBV (i.e. hepatitis B surface [HBs] antigen negative-, anti-HBs antibody positive and anti-hepatitis B core [HBc] antibody negative) or positive anti-HBc antibody from intravenous immunoglobulins (IVIG) may participate
* Treatment with any of the following within 7 days prior to the first dose of study drug:

  * Steroid therapy for anti-neoplastic intent
  * Moderate or strong cytochrome P450 3A (CYP3A) inhibitors
  * Moderate or strong CYP3A inducers
* Administration or consumption of any of the following within 3 days prior to the first dose of study drug:

  * Grapefruit or grapefruit products
  * Seville oranges (including marmalade containing Seville oranges)
  * Star fruit
* Patients with active hepatitis B infection (not including patients with prior hepatitis B vaccination; or positive serum hepatitis B antibody). Known hepatitis C infection is allowed as long as there is no active disease and is cleared by gastrointestinal (GI) consultation
* Central nervous system with mantle cell lymphoma
* Significant neuropathy (grades 3 to 4, or grade 2 with pain) within 14 days prior to enrollment
* Contraindication to any of the required concomitant drugs or supportive treatments or intolerance to hydration due to preexisting pulmonary or cardiac impairment including pleural effusion requiring thoracentesis or ascites requiring paracentesis unless due to lymphoma
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction, or any other gastrointestinal condition that could interfere with the absorption and metabolism of ibrutinib
* Major surgery within 4 weeks of initiation of therapy or a wound that has not fully healed within 4 weeks of randomization. Clearance letter from primary physician required
* Requires anticoagulation with warfarin or equivalent vitamin K antagonist
* Requires chronic treatment with strong CYP3A inhibitors
* Patients with New York Health Association (NYHA) Class III and IV heart failure, myocardial infarction in the preceding 6 months, and significant conduction abnormalities, including but not limited to left bundle branch block, 2nd degree atrioventricular (AV) block type II, 3rd degree block, QT prolongation (corrected QT [QTc] > 500 msec), sick sinus syndrome, ventricular tachycardia, symptomatic bradycardia (heart rate < 50 bpm), hypotension, light headedness and syncope, persistent and uncontrolled atrial fibrillation
* Recent placement of a stent and by recommendation of their cardiologist need to stay on anticoagulants such as warfarin or equivalent vitamin K antagonist
* Acute infection requiring treatment (IV antibiotics, antivirals, or antifungals) within 14 days prior to initiation of therapy
* Child-Pugh class B or C are excluded
* Vaccinated with live, attenuated vaccines within 4 weeks of randomization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2027-03-22 (Estimated); Study Completion 2027-03-22 (Estimated)

PRIMARY OUTCOMES:
Efficacy of ibrutinib plus rituximab combination followed by venetoclax | Up to cycle 12
  Determined by complete response (CR). The complete response after 4 cycles of venetoclax combined with ibrutinib plus rituximab and toxicity within first cycle of venetoclax combination will be monitored simultaneously using the Bayesian stopping boundaries calculated based on beta-binomial distributions. The prior probabilities of response and toxicity are modeled by beta distributions. Complete response and its 95% confidence interval will be calculated. Logistic regression will be utilized to assess the effect of patient prognostic factors on the CR rate and the toxicity rate.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 5 years
  Graded according to Common Terminology Criteria for Adverse Events (CTCAE). The safety is measured by toxicity which is defined as grade 3-4 non-hematologic toxicities within first cycle treatment of venetoclax combined with ibrutinib plus rituximab. Toxicity data by type and severity will be summarized by frequency tables. Logistic regression will be utilized to assess the effect of patient prognostic factors on the CR rate and the toxicity rate.
Progression-free survival (PFS) | Up to 5 years
  The distribution of PFS will be estimated using the method of Kaplan and Meier. Comparison of PFS by important subgroups will be made using the log-rank test.

OTHER OUTCOMES:
Circulating tumor deoxyribonucleic acid (ctDNA) levels | Up to 5 years
  Descriptive statistics will be used to summarize the ctDNA levels. Longitudinal analysis will be applied to evaluate the change of over time for each detected variant using mixed-effects model. Dynamic prediction modeling with time-dependent covariate in survival analysis for PFS will be explored based on ctDNA levels and clinical covariates.

CONTACTS AND LOCATIONS:
Overall Officials: Luhua (Michael) Wang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org